CLINICAL TRIAL: NCT06387758
Title: Low Systemic/High Local Exercise Load in Pediatric Sickle Cell Disease
Brief Title: Low Systemic/High Local Exercise Load in Peds SCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UMMC-IRB-2022-473
Record Dates: First submitted 2024-04-08; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Anemia in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low systemic strength training (Experimental): 8-week (3 times per week; 45-minute sessions) home-based telehealth strengthening exercise program
  Interventions: Behavioral: Low systemic strength training
- Moderate systemic exercise (Experimental): 8-week (3 times per week; 45-minute sessions) home-based telehealth walking protocol
  Interventions: Behavioral: Moderate systemic exercise

INTERVENTIONS:
Behavioral: Low systemic strength training — Low systemic strength training. Youth will complete exercise training for 45 minutes. Eight specific exercises will be performed to target all major muscle groups: calf raises, handgrip, squats, seated row, chest press, plank, low bac extension, and crunches (Table 1). Each exercise involves contractions with moderate load but with an extended duration of up to five minutes.16,17 During each exercise session, youth will have a 5-minute warm up, 5-minute cool down, and be allowed to take rest breaks as needed (minimum 30 seconds). Youth will initially progress by decreasing the number of rest periods and then increasing load. Youth will be provided a 2 lb medicine ball, resistance weight bands, Thera Putty, and a Yoga mat for home exercises. Youth will keep this home exercise equipment.
  Arms: Low systemic strength training
Behavioral: Moderate systemic exercise — Youth assigned to the moderate systemic exercise load group will perform whole-body aerobic exercise at 40-59% of heart rate reserve (HRR) for 45 minutes.76,111 Youth will complete moderate systemic aerobic exercise by walking at a brisk pace and swinging their arms as they walk. Exercise personnel will supervise a 5-minute warm up and 5-minute cool down via videoconferencing and remain on the phone with youth at all times during the walking exercise session. Youth will exercise until the prescribed duration is achieved or until fatigue at which point they will either reduce the intensity or stop until they recover. All training intensities will be based around HRR so it is individualized (not exceeding 59% of HRR). Youth unable to meet the initial training requirements will be slowly progressed over the 8 weeks.
  Arms: Moderate systemic exercise

SUMMARY:
This research study wants to learn about what kind of exercise is best for kids with sickle cell disease. Participating children will have a small amount of blood drawn one time at the beginning of the study. Children will then complete some questionnaires that measure pain, physical function, and emotions (depression, anxiety) and complete some tests that measure physical fitness at the beginning and end of the study. Children will be randomized to either a home-based telehealth (1) walking or (2) strengthening exercise program that lasts for 8-weeks, 3-x week, for 45 minutes each session. Children's participation will last up to 10 weeks.

DETAILED DESCRIPTION:
Overview: The current pilot study is a randomized behavioral exercise intervention.

Procedures:

Study Phase I: Families (n=60) will complete a baseline research visit. Youth will then be randomized to one of the exercise groups and complete one instructional exercise session, in person, at the UMMC Center for Integrative Health (CIH). After the instructional exercise session youth will complete a 3-day home ambulatory monitoring protocol. Study Phase II: Youth will then complete an 8-week Telehealth home exercise protocol. Youth will complete a 3-day ambulatory monitoring protocol during weeks 4 and 8. Youth will return to the UMMC CIH within one week of completing the exercise protocol to repeat questionnaires and clinical assessment. Parents will also repeat questionnaires.

Study Phase I:

Baseline Research Visit: Once enrolled, the RA will obtain parent contact information and contact information for two other relations. Youth and their parent will complete questionnaires using REDCap electronic data collection on Apple iPads (10 minutes). Questionnaires will include items on demographics, pain, physical functioning, and negative emotions (due to depression and negative affect being among the most robust predictors of pain in youth with SCD11,63,112,113). Blood draw: A blood sample will be collected (10 minutes) for the purpose of measuring baseline inflammatory markers. Every effort will be made to collect blood during scheduled clinical blood draws and using topical lidocaine cream. Clinical and Physical fitness assessment: Next, an Actigraph GT9X-BT device will be placed on youth's wrist to monitor HRV for the duration of the baseline research visit. Youth will then complete clinical and physical fitness assessments (30 minutes; detailed below).

Exercise Intervention: Randomization. Sixty numbers will be randomly assigned to either the low systemic strength training or the moderate systemic exercise groups in a 2:1 manner using the Microsoft Excel 2013 RANDBETWEEN1,2 function. Randomization order will be password protected and unlocked just prior to the instructional exercise session. However, of note, if families indicate that they do not have a safe environment to complete the moderate systemic exercise intervention (i.e., do not have a safe place to walk outside), then the youth participant will be assigned to the low systemic strength training group. The next eligible participant will be assigned to the moderate systemic exercise group to fulfill that randomization. Instructional Exercise Session. Youth will perform one 45-minute exercise session in-person at the UMMC CIH center. Prior to beginning exercise, exercise personnel will educate youth and parents regarding safe exercise (e.g., staying hydrated, moderate exercise levels) and potential adverse events75 (e.g., fatigue, muscle soreness; see Protections against risks, Exercise Sessions for more detail). At 5 minutes before exercise; 10, 20, 30, and 40 minutes during exercise, and 5 minutes after exercise pain intensity (primary outcome) and HRV (secondary outcome) will be obtained. 3-day Ambulatory Monitoring. Following the instructional exercise session, youth will partake in 3 consecutive days of actigraphy ambulatory monitoring and complete three days of pain diary. An actigraph is worn like a watch on the wrist of your non-dominant hand and measures physical activity, sleep, and heart-rate through light and movement and heartrate variability through a heart rate monitor. Daily diary pain intensity and actigraphy-derived HRV at 24-hours will be collected and contribute toward Aim 1: Hypotheses 1a and 1b. To reduce participant burden, wrist-worn Actigraphy devices will be returned via standard mail in a padded envelope.10

Study Phase II:

8-Week Telehealth Exercise Protocol. Using a within- and between-subject design, youth will serve as their own control (pre-post) and will complete 8-weeks (3 times per week; 45-minute sessions) of either (1) low systemic strength training or (2) moderate systemic exercise training. After the instructional exercise session, all exercise sessions will be completed at the home and supervised by study exercise personnel via Telehealth. A parent must also be present in the home during each exercise session. If a parent is not present, the exercise session will be rescheduled. Exercise personnel will record exercise adverse events at each session. All adverse events will be immediately reported to the medical director and PI.

3-day Ambulatory Monitoring. During week 4 and week 8 of the Telehealth exercise protocol, youth will partake in 3 consecutive days of daily diary and actigraphy ambulatory monitoring. Wrist-worn actigraphy devices will be returned via standard mail in a padded envelope and/or at the follow-up visit.

Follow-Up Visit. Families will return to the UMMC CIH within 1 week of completing the 8-week Telehealth exercise protocol. Youth will repeat questionnaires on pain (primary outcome, Aim 2) and assessment of HRV and physical fitness (secondary outcomes, Aim 2). Parents will also repeat questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* youth 12 to 17 years old
* diagnosed with SCD genotype SS, SC, beta-plus thalassemia, or beta-zero thalassemia
* has daily access to an Internet enabled device (e.g., smart phone, IPad) A parent (≥21 years old) will also be recruited for each youth participant.

Exclusion Criteria:

* non-English speaking due to lack of available written translation services for informed consent and questionnaires
* cognitive impairment (e.g., moderate to profound intellectual disability) that precludes study completion
* medical condition (e.g., hypertension, bone fracture) that precludes completing exercise safely (determined by study medical director Dr. McNaull).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Demographics and medical history (parents) | through study completion, an avg. of 10 weeks
  Parent name, address, email, social media contact information, child age, gender, diagnosis, prescribed medication dose and frequency, grade in school, parent marital status, parent education, and family income.
Pediatric Pain Questionnaire | through study completion, an avg. of 10 weeks
  The Pediatric Pain Questionnaire (PPQ, youth and parent version) is well-validated and consists of two 100 mm visual analogue scale items that measure present pain intensity and worst pain in the past week. One question of pain frequency will be added (0 = not at all to 6 = daily pain). The present pain intensity item will measure pain intensity during exercise sessions.
Functional Disability Inventory | through study completion, an avg. of 10 weeks
  The Functional Disability Inventory (FDI, youth and parent version)79 is a 15-item well-validated scale assessing difficulty in physical and psychosocial functioning due to physical health (0 = no trouble to 4 = impossible).80,81
NIH PROMIS 2582 | through study completion, an avg. of 10 weeks
  The NIH PROMIS 2582 (youth and parent-proxy) includes 25-items on physical function mobility, anxiety, depression, fatigue, peer relations, pain interference, and pain intensity. Items are scored on a 5-point Likert scale and converted to standard T-scores; except pain intensity (10-point numeric rating scale).
Heart Rate Variability | through study completion, an avg. of 10 weeks
  HRV for both Phase I and II will be recorded using the Actigraph GT9X-BT device capable of collecting R-R intervals, and in accordance with established guidelines.22 Time Domain measures will include the standard deviation of normal RR intervals (SDNN, reflects sympathetic activity), and the square root of the mean squared differences between normal adjacent R-R intervals (RMSSD, reflects parasympathetic activity). Spectral analysis of HRV will be derived via a 1024-point linear fast Fourier transformation using a Hamming window. The resultant power density spectrum will be analyzed for total power (0.00-0.40 Hz), LF (0.04-0.15 Hz), and HF (0.15-0.40 Hz). LF and HF will be further normalized (LFNU and HFNU) to quantify sympathovagal balance.
Heart Rate | through study completion, an avg. of 10 weeks
  Vital Signs measured will include heart rate (Phillips Healthcare; Netherlands).
Blood Pressure | through study completion, an avg. of 10 weeks
  Vital Signs measured will include blood pressure (BP). Systolic and diastolic blood pressure will be measured following a 5-minute rest period, three times (1 minute apart) in the non-dominant arm using automated oscillometric measurement and an appropriate-sized cuff.
Bruininks-Oseretsky Test of Motor Proficiency | through study completion, an avg. of 10 weeks
  Physical fitness will be assessed using the well-validated Bruininks-Oseretsky Test of Motor Proficiency, 2nd edition (4-21 years) to measure upper-limb and bilateral coordination, balance, running speed and agility, and strength.86,87 Aerobic endurance will be measured using American Thoracic Society 6-minute walk test guidelines. Dr. Daniels will train exercise personnel and the study RA in clinical assessment to proficiency and review 30% of data for research fidelity.
American Thoracic Society 6-minute walk test | through study completion, an avg. of 10 weeks
  Aerobic endurance will be measured using American Thoracic Society 6-minute walk test guidelines. Dr. Daniels will train exercise personnel and the study RA in clinical assessment to proficiency and review 30% of data for research fidelity.
Actigraphy | through study completion, an avg. of 10 weeks
  Objective recordings of daily HRV will be assessed with an Actigraph GT9X-BT device and computed using the ActiLife 6 software package. The watch-like device is worn on the non-dominant wrist.92 Wrist actigraphy has been validated in both healthy children and children with chronic pain.92-95
Daily diaries | through study completion, an avg. of 10 weeks
  Diary items are derived from the above questionnaires, created in REDCap, take less than 3 minutes to answer, and will be completed once in the evening at a specified time. A diary link will be texted or emailed to the participant's smartphone or computer. Diary items will include: pain duration (pain start and stop time), pain intensity (100 mm visual analogue scale), daily mood (e.g., worried, sad), pain medications, and functional disability. All diary information will be immediately encrypted in REDCap.
Biomarkers | pre- 2 weeks
  Utilizing the UMMC Immunology Biomarker Core under senior mentor Dr. Marshall, we will measure inflammatory IL-6, TNF-α, and CRP biomarker18-21 levels. 10 mL whole blood samples will be collected in heparinized tubes.96-98 Plasma samples will be rapidly obtained by centrifugation and will be stored at -80◦C in a research freezer until batch analyzed. Inflammatory marker IL-6 and TNF-α concentrations will be analyzed using Luminex® assay kits. We will examine CRP and using antibody-sandwich ELISA (Assaypro LLC, St. Charles, MO). Standard laboratory and assay measurement limits, normal and cut-off age values will be used to define absolute and high values.
Medical Chart Review | pre- 2 weeks
  The following variables will be extracted from youth's electronic health record: date of birth, diagnoses, prescribed medications, complications, blood laboratory results over the past year, height and weight at last clinic visits, and number of emergency room visits and hospitalizations for pain during past three years. Complications and pain-related visits/hospitalizations will determine SCD disease severity. A potential concern in this study is the broad age range of 12-17 year olds, with children's changing immune system and differences in pubertal Tanner stage potentially impacting their physiological response to exercise. Thus, age and estimated pubertal Tanner stage will be examined as possible covariates. Pubertal status according to Tanner Stage criteria will be estimated by the pediatric hematologist/nurse practitioner at a regular office visit. All practitioners have appropriate training in pediatric examination.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Griffin, Study Director — Director-Clinical Trials Office
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available from researchers upon reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years after study completion/publication
Access Criteria: Email communication

REFERENCES:
- [Background] Steinberg MH. Sickle cell anemia, the first molecular disease: overview of molecular etiology, pathophysiology, and therapeutic approaches. ScientificWorldJournal. 2008 Dec 25;8:1295-324. doi: 10.1100/tsw.2008.157. PMID 19112541
- [Background] Piel FB, Patil AP, Howes RE, Nyangiri OA, Gething PW, Dewi M, Temperley WH, Williams TN, Weatherall DJ, Hay SI. Global epidemiology of sickle haemoglobin in neonates: a contemporary geostatistical model-based map and population estimates. Lancet. 2013 Jan 12;381(9861):142-51. doi: 10.1016/S0140-6736(12)61229-X. Epub 2012 Oct 25. PMID 23103089
- [Background] Cooper L, Walker T, Polk B, Smith L, Karlson C, Rhodes M, Majumdar S. Estimate and cost of hemoglobin disorders among African Americans in Mississippi. Journal for Mississippi State Medical Association. 2018.
- [Background] Sil S, Cohen LL, Dampier C. Psychosocial and Functional Outcomes in Youth With Chronic Sickle Cell Pain. Clin J Pain. 2016 Jun;32(6):527-33. doi: 10.1097/AJP.0000000000000289. PMID 26379074
- [Background] Kuntze G, Nesbitt C, Whittaker JL, Nettel-Aguirre A, Toomey C, Esau S, Doyle-Baker PK, Shank J, Brooks J, Benseler S, Emery CA. Exercise Therapy in Juvenile Idiopathic Arthritis: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Jan;99(1):178-193.e1. doi: 10.1016/j.apmr.2017.05.030. Epub 2017 Jul 18. PMID 28729171
- [Background] Dougherty KA, Bertolaso C, Schall JI, Smith-Whitley K, Stallings VA. Muscle Strength, Power, and Torque Deficits in Children With Type SS Sickle Cell Disease. J Pediatr Hematol Oncol. 2018 Jul;40(5):348-354. doi: 10.1097/MPH.0000000000001143. PMID 29621064
- [Background] Martin C, Pialoux V, Faes C, Charrin E, Skinner S, Connes P. Does physical activity increase or decrease the risk of sickle cell disease complications? Br J Sports Med. 2018 Feb;52(4):214-218. doi: 10.1136/bjsports-2015-095317. Epub 2015 Dec 23. PMID 26701924
- [Background] Merlet AN, Chatel B, Hourde C, Ravelojaona M, Bendahan D, Feasson L, Messonnier LA. How Sickle Cell Disease Impairs Skeletal Muscle Function: Implications in Daily Life. Med Sci Sports Exerc. 2019 Jan;51(1):4-11. doi: 10.1249/MSS.0000000000001757. PMID 30095751
- [Background] National Institutes of Health, National Heart, Lung, and Blood Institute, Division of Blood Diseases and Resources. The management of sickle cell disease (NIH publication no. 02-2117). 2002 Jun. Available from: http://www.nhlbi.nih.gov/files/docs/guidelines/sc_mngt.pdf.
- [Background] Karlson CW, Baker AM, Bromberg MH, David Elkin T, Majumdar S, Palermo TM. Daily Pain, Physical Activity, and Home Fluid Intake in Pediatric Sickle Cell Disease. J Pediatr Psychol. 2017 Apr 1;42(3):335-344. doi: 10.1093/jpepsy/jsw061. PMID 27370016
- [Background] Karlson CW, Delozier AM, Seals SR, Britt AB, Stone AL, Reneker JC, Jackson EA, McNaull MM, Credeur DP, Welsch MA. Physical Activity and Pain in Youth With Sickle Cell Disease. Fam Community Health. 2020 Jan/Mar;43(1):1-9. doi: 10.1097/FCH.0000000000000241. PMID 31764301
- [Background] Badawy SM, Payne AB, Rodeghier MJ, Liem RI. Exercise capacity and clinical outcomes in adults followed in the Cooperative Study of Sickle Cell Disease (CSSCD). Eur J Haematol. 2018 Oct;101(4):532-541. doi: 10.1111/ejh.13140. Epub 2018 Aug 31. PMID 29999202
- [Background] Abd El-Kader SM, Al-Shreef FM. Impact of aerobic exercises on selected inflammatory markers and immune system response among patients with sickle cell anemia in asymptomatic steady state. Afr Health Sci. 2018 Mar;18(1):111-119. doi: 10.4314/ahs.v18i1.15. PMID 29977264
- [Background] Gellen B, Messonnier LA, Galacteros F, Audureau E, Merlet AN, Rupp T, Peyrot S, Martin C, Feasson L, Bartolucci P; EXDRE collaborative study group. Moderate-intensity endurance-exercise training in patients with sickle-cell disease without severe chronic complications (EXDRE): an open-label randomised controlled trial. Lancet Haematol. 2018 Nov;5(11):e554-e562. doi: 10.1016/S2352-3026(18)30163-7. PMID 30389037
- [Background] Liem RI, Akinosun M, Muntz DS, Thompson AA. Feasibility and safety of home exercise training in children with sickle cell anemia. Pediatr Blood Cancer. 2017 Dec;64(12). doi: 10.1002/pbc.26671. Epub 2017 Jun 9. PMID 28598539
- [Background] Allen JD, Robbins JL, Vanbruggen MD, Credeur DP, Johannsen NM, Earnest CP, Pieper CF, Johnson JL, Church TS, Ravussin E, Kraus WE, Welsch MA. Unlocking the barriers to improved functional capacity in the elderly: rationale and design for the "Fit for Life trial". Contemp Clin Trials. 2013 Sep;36(1):266-75. doi: 10.1016/j.cct.2013.07.007. Epub 2013 Jul 27. PMID 23900005
- [Background] Allen JD, Vanbruggen MD, Johannsen NM, Robbins JL, Credeur DP, Pieper CF, Sloane R, Earnest CP, Church TS, Ravussin E, Kraus WE, Welsch MA. PRIME: A Novel Low-Mass, High-Repetition Approach to Improve Function in Older Adults. Med Sci Sports Exerc. 2018 May;50(5):1005-1014. doi: 10.1249/MSS.0000000000001518. PMID 29232316
- [Background] Belcher JD, Mahaseth H, Welch TE, Vilback AE, Sonbol KM, Kalambur VS, Bowlin PR, Bischof JC, Hebbel RP, Vercellotti GM. Critical role of endothelial cell activation in hypoxia-induced vasoocclusion in transgenic sickle mice. Am J Physiol Heart Circ Physiol. 2005 Jun;288(6):H2715-25. doi: 10.1152/ajpheart.00986.2004. Epub 2005 Jan 21. PMID 15665055
- [Background] Krishnan S, Setty Y, Betal SG, Vijender V, Rao K, Dampier C, Stuart M. Increased levels of the inflammatory biomarker C-reactive protein at baseline are associated with childhood sickle cell vasocclusive crises. Br J Haematol. 2010 Mar;148(5):797-804. doi: 10.1111/j.1365-2141.2009.08013.x. Epub 2009 Dec 8. PMID 19995398
- [Background] Platt OS. Sickle cell anemia as an inflammatory disease. J Clin Invest. 2000 Aug;106(3):337-8. doi: 10.1172/JCI10726. No abstract available. PMID 10930436
- [Background] Sarray S, Saleh LR, Lisa Saldanha F, Al-Habboubi HH, Mahdi N, Almawi WY. Serum IL-6, IL-10, and TNFalpha levels in pediatric sickle cell disease patients during vasoocclusive crisis and steady state condition. Cytokine. 2015 Mar;72(1):43-7. doi: 10.1016/j.cyto.2014.11.030. Epub 2015 Jan 5. PMID 25569375
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Wood RH, Wood WA, Welsch M, Avenal P. Physical activity, mental stress, and short-term heart rate variability in patients with ischemic heart disease. J Cardiopulm Rehabil. 1998 Jul-Aug;18(4):271-6. doi: 10.1097/00008483-199807000-00003. PMID 9702605
- [Background] Kluess HA, Wood RH, Welsch MA. Vagal modulation of the heart and central hemodynamics during handgrip exercise. Am J Physiol Heart Circ Physiol. 2000 May;278(5):H1648-52. doi: 10.1152/ajpheart.2000.278.5.H1648. PMID 10775145
- [Background] Lee CM, Aucoin NA, Wood RH, Welsch MA, Kalb D. Short-term heart rate variability in type-I diabetics: the influence of breathing pattern and exercise capacity. Clinical Exercise Physiology. 2 (2):72-76, 2000.
- [Background] Lee CM, Wood RH, Welsch MA. Influence of head-down and lateral decubitus neck flexion on heart rate variability. J Appl Physiol (1985). 2001 Jan;90(1):127-32. doi: 10.1152/jappl.2001.90.1.127. PMID 11133902
- [Background] Wood RH, Leleux S, Welsch MA, Nelson AG, Lee AM. Heart rate variability following 5 weeks of detraining in competitive swimmers. Medicina Standiva 5 (1) pp. E49-E58, 2001.
- [Background] Lee CM, Wood RH, Welsch MA. Influence of short-term endurance exercise training on heart rate variability. Med Sci Sports Exerc. 2003 Jun;35(6):961-9. doi: 10.1249/01.MSS.0000069410.56710.DA. PMID 12783044
- [Background] Dos Santos JP, Gomes Neto M. Sociodemographic aspects and quality of life of patients with sickle cell anemia. Rev Bras Hematol Hemoter. 2013;35(4):242-5. doi: 10.5581/1516-8484.20130093. PMID 24106440
- [Background] Sil S, Cohen LL, Dampier C. Pediatric pain screening identifies youth at risk of chronic pain in sickle cell disease. Pediatr Blood Cancer. 2019 Mar;66(3):e27538. doi: 10.1002/pbc.27538. Epub 2018 Nov 4. PMID 30393948
- [Background] Ladd RJ, Valrie CR, Walcott CM. Risk and resilience factors for grade retention in youth with sickle cell disease. Pediatr Blood Cancer. 2014 Jul;61(7):1252-6. doi: 10.1002/pbc.24974. Epub 2014 Feb 12. PMID 24519984
- [Background] Aljuburi G, Laverty AA, Green SA, Phekoo KJ, Bell D, Majeed A. Socio-economic deprivation and risk of emergency readmission and inpatient mortality in people with sickle cell disease in England: observational study. J Public Health (Oxf). 2013 Dec;35(4):510-7. doi: 10.1093/pubmed/fdt100. Epub 2013 Oct 29. PMID 24169414
- [Background] Asnani MR, Knight Madden J, Reid M, Greene LG, Lyew-Ayee P. Socio-environmental exposures and health outcomes among persons with sickle cell disease. PLoS One. 2017 Apr 6;12(4):e0175260. doi: 10.1371/journal.pone.0175260. eCollection 2017. PMID 28384224
- [Background] Robinson MR, Daniel LC, O'Hara EA, Szabo MM, Barakat LP. Insurance status as a sociodemographic risk factor for functional outcomes and health-related quality of life among youth with sickle cell disease. J Pediatr Hematol Oncol. 2014 Jan;36(1):51-6. doi: 10.1097/MPH.0000000000000013. PMID 24136028
- [Background] Syrop J. Bill addressing sickle cell disease/heritable blood disorders signed into law. [Internet]. AJMC. 2018 Dec 29. Available from: https://www.ajmc.com/newsroom/bill-addressing-sickle-cell-diseaseheritable-blood-disorders-signed-into-law
- [Background] Strouse JJ, Lobner K, Lanzkron S, MHS, Haywood C Jr. NIH and national foundation expenditures for sickle cell disease and cystic fibrosis are associated with Pubmed publications and FDA approvals. Blood 2013:122:1739.
- [Background] Dampier C, Palermo TM, Darbari DS, Hassell K, Smith W, Zempsky W. AAPT Diagnostic Criteria for Chronic Sickle Cell Disease Pain. J Pain. 2017 May;18(5):490-498. doi: 10.1016/j.jpain.2016.12.016. Epub 2017 Jan 5. PMID 28065813
- [Background] Han J, Zhou J, Saraf SL, Gordeuk VR, Calip GS. Characterization of opioid use in sickle cell disease. Pharmacoepidemiol Drug Saf. 2018 May;27(5):479-486. doi: 10.1002/pds.4291. Epub 2017 Aug 16. PMID 28815799
- [Background] National Institutes of Health, National Heart, Lung, and Blood Institute. Evidence-Based Management of Sickle Cell Disease: Expert Panel Report, 2014. (Report. 020816_0). 2014 Sep. Available from: http://www.nhlbi.nih.gov/guidelines.
- [Background] Steinberg MH. Management of sickle cell disease. N Engl J Med. 1999 Apr 1;340(13):1021-30. doi: 10.1056/NEJM199904013401307. No abstract available. PMID 10099145
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Hojsted J, Kurita GP, Kendall S, Lundorff L, de Mattos Pimenta CA, Sjogren P. Non-analgesic effects of opioids: the cognitive effects of opioids in chronic pain of malignant and non-malignant origin. An update. Curr Pharm Des. 2012;18(37):6116-22. doi: 10.2174/138161212803582522. PMID 22747540
- [Background] Fearon A, Marsh A, Kim J, Treadwell M. Pediatric residents' perceived barriers to opioid use in sickle cell disease pain management. Pediatr Blood Cancer. 2019 Feb;66(2):e27535. doi: 10.1002/pbc.27535. Epub 2018 Nov 1. PMID 30387290
- [Background] Feliu MH, Wellington C, Crawford RD, Wood M, Edwards L, Byrd G, Edwards CL. Opioid management and dependency among adult patients with sickle cell disease. Hemoglobin. 2011;35(5-6):485-94. doi: 10.3109/03630269.2011.610914. Epub 2011 Sep 12. PMID 21910605
- [Background] Hechler T, Kanstrup M, Holley AL, Simons LE, Wicksell R, Hirschfeld G, Zernikow B. Systematic Review on Intensive Interdisciplinary Pain Treatment of Children With Chronic Pain. Pediatrics. 2015 Jul;136(1):115-27. doi: 10.1542/peds.2014-3319. Epub 2015 Jun 22. PMID 26101358
- [Background] Pearson SR, Alkon A, Treadwell M, Wolff B, Quirolo K, Boyce WT. Autonomic reactivity and clinical severity in children with sickle cell disease. Clin Auton Res. 2005 Dec;15(6):400-7. doi: 10.1007/s10286-005-0300-9. PMID 16362543
- [Background] Connes P, Machado R, Hue O, Reid H. Exercise limitation, exercise testing and exercise recommendations in sickle cell anemia. Clin Hemorheol Microcirc. 2011;49(1-4):151-63. doi: 10.3233/CH-2011-1465. PMID 22214686
- [Background] Tewari S, Brousse V, Piel FB, Menzel S, Rees DC. Environmental determinants of severity in sickle cell disease. Haematologica. 2015 Sep;100(9):1108-16. doi: 10.3324/haematol.2014.120030. PMID 26341524
- [Background] Chatel B, Messonnier LA, Barge Q, Vilmen C, Noirez P, Bernard M, Pialoux V, Bendahan D. Endurance training reduces exercise-induced acidosis and improves muscle function in a mouse model of sickle cell disease. Mol Genet Metab. 2018 Mar;123(3):400-410. doi: 10.1016/j.ymgme.2017.11.010. Epub 2017 Nov 28. PMID 29307759
- [Background] Neumayr LD, Aguilar C, Earles AN, Jergesen HE, Haberkern CM, Kammen BF, Nancarrow PA, Padua E, Milet M, Stulberg BN, Williams RA, Orringer EP, Graber N, Robertson SM, Vichinsky EP; National Osteonecrosis Trial in Sickle Cell Anemia Study Group. Physical therapy alone compared with core decompression and physical therapy for femoral head osteonecrosis in sickle cell disease. Results of a multicenter study at a mean of three years after treatment. J Bone Joint Surg Am. 2006 Dec;88(12):2573-82. doi: 10.2106/JBJS.E.01454. PMID 17142406
- [Background] Coimbra S, Catarino C, Nascimento H, Ines Alves A, Filipa Medeiros A, Bronze-da-Rocha E, Costa E, Rocha-Pereira P, Aires L, Seabra A, Mota J, Ferreira Mansilha H, Rego C, Santos-Silva A, Belo L. Physical exercise intervention at school improved hepcidin, inflammation, and iron metabolism in overweight and obese children and adolescents. Pediatr Res. 2017 Nov;82(5):781-788. doi: 10.1038/pr.2017.139. Epub 2017 Jul 19. PMID 28604755
- [Background] Remmel L, Tillmann V, Mengel E, Kool P, Purge P, Latt E, Jurimae J. The Impact of Physical Activity on Serum Inflammatory Markers in Overweight Pubertal Boys: 24-Month Follow-Up Study. Pediatr Exerc Sci. 2018 May 1;30(2):198-207. doi: 10.1123/pes.2016-0252. Epub 2017 Dec 23. PMID 29276854
- [Background] Sloan RP, Shapiro PA, McKinley PS, Bartels M, Shimbo D, Lauriola V, Karmally W, Pavlicova M, Choi CJ, Choo TH, Scodes JM, Flood P, Tracey KJ. Aerobic Exercise Training and Inducible Inflammation: Results of a Randomized Controlled Trial in Healthy, Young Adults. J Am Heart Assoc. 2018 Sep 4;7(17):e010201. doi: 10.1161/JAHA.118.010201. PMID 30371169
- [Background] Baker AM, Raiker JS, Elkin TD, Palermo TM, Karlson CW. Internalizing symptoms mediate the relationship between sleep disordered breathing and pain symptoms in a pediatric hematology/oncology sample. Children's Health Care. 2017:46:34-48. doi: 10.1080/02739615.2015.1124326
- [Background] Fisher K, Laikin AM, Sharp KMH, Criddle CA, Palermo TM, Karlson CW. Temporal relationship between daily pain and actigraphy sleep patterns in pediatric sickle cell disease. J Behav Med. 2018 Jun;41(3):416-422. doi: 10.1007/s10865-018-9918-7. Epub 2018 Mar 12. PMID 29532199
- [Background] Lim CS, Karlson C, Edmond SN, Welkom JS, Osunkwo I, Cohen LL. Emotion-Focused Avoidance Coping Mediates the Association Between Pain and Health-Related Quality of Life in Children With Sickle Cell Disease. J Pediatr Hematol Oncol. 2019 Apr;41(3):194-201. doi: 10.1097/MPH.0000000000001429. PMID 30720675
- [Background] Karlson CW, Leist-Haynes S, Smith M, Faith MA, Elkin TD, Megason G. Examination of risk and resiliency in a pediatric sickle cell disease population using the psychosocial assessment tool 2.0. J Pediatr Psychol. 2012 Oct;37(9):1031-40. doi: 10.1093/jpepsy/jss087. Epub 2012 Jul 26. PMID 22836746
- [Background] Palermo TM, Valrie CR, Karlson CW. Family and parent influences on pediatric chronic pain: a developmental perspective. Am Psychol. 2014 Feb-Mar;69(2):142-52. doi: 10.1037/a0035216. PMID 24547800
- [Background] Rabbitts JA, Holley AL, Karlson CW, Palermo TM. Bidirectional associations between pain and physical activity in adolescents. Clin J Pain. 2014 Mar;30(3):251-8. doi: 10.1097/AJP.0b013e31829550c6. PMID 23669450
- [Background] Rapoff MA, Connelly M, Bickel JL, Powers SW, Hershey AD, Allen JR, Karlson CW, Litzenburg CC, Belmont JM. Headstrong intervention for pediatric migraine headache: a randomized clinical trial. J Headache Pain. 2014 Feb 28;15(1):12. doi: 10.1186/1129-2377-15-12. PMID 24580721
- [Background] Stone AL, Karlson CW, Heathcote LC, Rosenberg AR, Palermo TM. Topical Review: Pain in Survivors of Pediatric Cancer: Applying a Prevention Framework. J Pediatr Psychol. 2018 Apr 1;43(3):237-242. doi: 10.1093/jpepsy/jsx114. PMID 29048571
- [Background] Alomari MA, Keewan EF, Shammaa RA, Alawneh K, Khatib SY, Welsch MA. Vascular function and handgrip strength in rheumatoid arthritis patients. ScientificWorldJournal. 2012;2012:580863. doi: 10.1100/2012/580863. Epub 2012 Mar 12. PMID 22606051
- [Background] Credeur DP, Dobrosielski DA, Arce-Esquivel AA, Welsch MA. Brachial artery retrograde flow increases with age: relationship to physical function. Eur J Appl Physiol. 2009 Sep;107(2):219-25. doi: 10.1007/s00421-009-1117-3. Epub 2009 Jun 30. PMID 19565260
- [Background] Credeur DP, Hollis BC, Welsch MA. Effects of handgrip training with venous restriction on brachial artery vasodilation. Med Sci Sports Exerc. 2010 Jul;42(7):1296-302. doi: 10.1249/MSS.0b013e3181ca7b06. PMID 20019641
- [Background] Credeur DP, Mariappan N, Francis J, Thomas D, Moraes D, Welsch MA. Vasoreactivity before and after handgrip training in chronic heart failure patients. Atherosclerosis. 2012 Nov;225(1):154-9. doi: 10.1016/j.atherosclerosis.2012.08.013. Epub 2012 Sep 16. PMID 23010159
- [Background] Godawa TM, Credeur DP, Welsch MA. Influence of compressive gear on powerlifting performance: role of blood flow restriction training. J Strength Cond Res. 2012 May;26(5):1274-80. doi: 10.1519/JSC.0b013e3182510643. PMID 22395280
- [Background] Welsch MA, Alomari M, Parish TR, Wood RH, Kalb D. Influence of venous function on exercise tolerance in chronic heart failure. J Cardiopulm Rehabil. 2002 Sep-Oct;22(5):321-6. doi: 10.1097/00008483-200209000-00002. PMID 12370591
- [Background] Welsch MA, Blalock P, Credeur DP, Parish TR. Comparison of brachial artery vasoreactivity in elite power athletes and age-matched controls. PLoS One. 2013;8(1):e54718. doi: 10.1371/journal.pone.0054718. Epub 2013 Jan 24. PMID 23359214
- [Background] Welsch MA, Pollock ML. Exercise Benefits and Prescription in Chronic Heart Failure: The Elderly Patient. Am J Geriatr Cardiol. 1996 Jan;5(1):71-77. No abstract available. PMID 11416371
- [Background] Dampier C, Ely B, Brodecki D, O'Neal P. Characteristics of pain managed at home in children and adolescents with sickle cell disease by using diary self-reports. J Pain. 2002 Dec;3(6):461-70. doi: 10.1054/jpai.2002.128064. PMID 14622732
- [Background] Stone AL, Williams Z, McNaull M, Wilson AC, Karlson CW. Daily Associations between Child and Parent Psychological Factors and Home Opioid Use in Youth with Sickle Cell Disease. Ann Behav Med. 2020 Jan 1;54(1):61-66. doi: 10.1093/abm/kaz022. PMID 31731289
- [Background] Burkhart PV, Dunbar-Jacob JM, Rohay JM. Accuracy of children's self-reported adherence to treatment. J Nurs Scholarsh. 2001;33(1):27-32. doi: 10.1111/j.1547-5069.2001.00027.x. PMID 11253577
- [Background] Carlesso LC, Macdermid JC, Santaguida LP. Standardization of adverse event terminology and reporting in orthopaedic physical therapy: application to the cervical spine. J Orthop Sports Phys Ther. 2010 Aug;40(8):455-63. doi: 10.2519/jospt.2010.3229. PMID 20710083
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Varni JW, Burwinkle TM, Katz ER. The PedsQL in pediatric cancer pain: a prospective longitudinal analysis of pain and emotional distress. J Dev Behav Pediatr. 2004 Aug;25(4):239-46. doi: 10.1097/00004703-200408000-00003. PMID 15308924
- [Background] Wilson AC, Palermo TM. Physical activity and function in adolescents with chronic pain: a controlled study using actigraphy. J Pain. 2012 Feb;13(2):121-30. doi: 10.1016/j.jpain.2011.08.008. Epub 2011 Nov 17. PMID 22099608
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Kashikar-Zuck S, Flowers SR, Claar RL, Guite JW, Logan DE, Lynch-Jordan AM, Palermo TM, Wilson AC. Clinical utility and validity of the Functional Disability Inventory among a multicenter sample of youth with chronic pain. Pain. 2011 Jul;152(7):1600-1607. doi: 10.1016/j.pain.2011.02.050. Epub 2011 Mar 31. PMID 21458162
- [Background] Claar RL, Walker LS. Functional assessment of pediatric pain patients: psychometric properties of the functional disability inventory. Pain. 2006 Mar;121(1-2):77-84. doi: 10.1016/j.pain.2005.12.002. Epub 2006 Feb 9. PMID 16480823
- [Background] Forrest CB, Bevans KB, Tucker C, Riley AW, Ravens-Sieberer U, Gardner W, Pajer K. Commentary: the patient-reported outcome measurement information system (PROMIS(R)) for children and youth: application to pediatric psychology. J Pediatr Psychol. 2012 Jul;37(6):614-21. doi: 10.1093/jpepsy/jss038. Epub 2012 Feb 23. No abstract available. PMID 22362923
- [Background] Pikilidou M, Yavropoulou M, Antoniou M, Papakonstantinou E, Pantelidou D, Chalkia P, Nilsson P, Yovos J, Zebekakis P. Arterial Stiffness and Peripheral and Central Blood Pressure in Patients With Sickle Cell Disease. J Clin Hypertens (Greenwich). 2015 Sep;17(9):726-31. doi: 10.1111/jch.12572. Epub 2015 May 20. PMID 25991400
- [Background] Negroni-Balasquide X, Bell CS, Samuel J, Samuels JA. Is one measurement enough to evaluate blood pressure among adolescents? A blood pressure screening experience in more than 9000 children with a subset comparison of auscultatory to mercury measurements. J Am Soc Hypertens. 2016 Feb;10(2):95-100. doi: 10.1016/j.jash.2015.12.001. Epub 2015 Dec 15. PMID 26875474
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Background] Gentier I, D'Hondt E, Shultz S, Deforche B, Augustijn M, Hoorne S, Verlaecke K, De Bourdeaudhuij I, Lenoir M. Fine and gross motor skills differ between healthy-weight and obese children. Res Dev Disabil. 2013 Nov;34(11):4043-51. doi: 10.1016/j.ridd.2013.08.040. Epub 2013 Sep 13. PMID 24036485
- [Background] Wali YA, Moheeb H. Effect of hydroxyurea on physical fitness indices in children with sickle cell anemia. Pediatr Hematol Oncol. 2011 Feb;28(1):43-50. doi: 10.3109/08880018.2010.524278. Epub 2010 Nov 17. PMID 21083357
- [Background] Agha H, El Tagui M, El Ghamrawy M, Abdel Hady M. The 6-min walk test: an independent correlate of elevated tricuspid regurgitant jet velocity in children and young adult sickle cell patients. Ann Hematol. 2014 Jul;93(7):1131-8. doi: 10.1007/s00277-014-2030-3. Epub 2014 Feb 22. PMID 24562420
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Finan PH, Carroll CP, Moscou-Jackson G, Martel MO, Campbell CM, Pressman A, Smyth JM, Tremblay JM, Lanzkron SM, Haythornthwaite JA. Daily Opioid Use Fluctuates as a Function of Pain, Catastrophizing, and Affect in Patients With Sickle Cell Disease: An Electronic Daily Diary Analysis. J Pain. 2018 Jan;19(1):46-56. doi: 10.1016/j.jpain.2017.08.010. Epub 2017 Sep 21. PMID 28943232
- [Background] Fine PG, Portenoy RK. A Clinical Guide to Opioid Analgesia. Minneapolis, MN: McGraw-Hill; 2004. Healthcare information programs.
- [Background] Ekblom O, Nyberg G, Bak EE, Ekelund U, Marcus C. Validity and comparability of a wrist-worn accelerometer in children. J Phys Act Health. 2012 Mar;9(3):389-93. PMID 22454440
- [Background] Kashikar-Zuck S, Flowers SR, Verkamp E, Ting TV, Lynch-Jordan AM, Graham TB, Passo M, Schikler KN, Hashkes PJ, Spalding S, Banez G, Richards MM, Powers SW, Arnold LM, Lovell D. Actigraphy-based physical activity monitoring in adolescents with juvenile primary fibromyalgia syndrome. J Pain. 2010 Sep;11(9):885-93. doi: 10.1016/j.jpain.2009.12.009. Epub 2010 Apr 24. PMID 20418183
- [Background] Long AC, Palermo TM, Manees AM. Brief report: using actigraphy to compare physical activity levels in adolescents with chronic pain and healthy adolescents. J Pediatr Psychol. 2008 Jul;33(6):660-5. doi: 10.1093/jpepsy/jsm136. Epub 2008 Jan 7. PMID 18180253
- [Background] Puyau MR, Adolph AL, Vohra FA, Butte NF. Validation and calibration of physical activity monitors in children. Obes Res. 2002 Mar;10(3):150-7. doi: 10.1038/oby.2002.24. PMID 11886937
- [Background] Heffner KL, Ng HM, Suhr JA, France CR, Marshall GD, Pigeon WR, Moynihan JA. Sleep disturbance and older adults' inflammatory responses to acute stress. Am J Geriatr Psychiatry. 2012 Sep;20(9):744-52. doi: 10.1097/JGP.0b013e31824361de. PMID 22327621
- [Background] Human IL-6 Platinum ELISA BMS213/2 / BMS213/2TEN: Enzyme-linked Immunosorbent Assay for quantitative detection of human IL-6. eBioscience. Accessed from www.eBioscience.com on November 4, 2016.
- [Background] Glaser R, Padgett DA, Litsky ML, Baiocchi RA, Yang EV, Chen M, Yeh PE, Klimas NG, Marshall GD, Whiteside T, Herberman R, Kiecolt-Glaser J, Williams MV. Stress-associated changes in the steady-state expression of latent Epstein-Barr virus: implications for chronic fatigue syndrome and cancer. Brain Behav Immun. 2005 Mar;19(2):91-103. doi: 10.1016/j.bbi.2004.09.001. PMID 15664781
- [Background] Hardy SJ, Bills SE, Wise SM, Hardy KK. Cognitive Abilities Moderate the Effect of Disease Severity on Health-Related Quality of Life in Pediatric Sickle Cell Disease. J Pediatr Psychol. 2018 Sep 1;43(8):882-894. doi: 10.1093/jpepsy/jsy019. PMID 29659914
- [Background] Tanner JM, Davies PS. Clinical longitudinal standards for height and height velocity for North American children. J Pediatr. 1985 Sep;107(3):317-29. doi: 10.1016/s0022-3476(85)80501-1. PMID 3875704
- [Background] Karlson CW, Rapoff MA. Attrition in randomized controlled trials for pediatric chronic conditions. J Pediatr Psychol. 2009 Aug;34(7):782-93. doi: 10.1093/jpepsy/jsn122. Epub 2008 Dec 8. PMID 19064607
- [Background] Tabachnick BG, Fidell LS. Using Multivariate Statistics. 5th rev. ed. Boston: Allyn and Bacon; 2007.
- [Background] Pediatric OCD Treatment Study (POTS) Team. Cognitive-behavior therapy, sertraline, and their combination for children and adolescents with obsessive-compulsive disorder: the Pediatric OCD Treatment Study (POTS) randomized controlled trial. JAMA. 2004 Oct 27;292(16):1969-76. doi: 10.1001/jama.292.16.1969. PMID 15507582
- [Background] Muthen LK, Muthen BO. User's guide. Los Angeles: Muthen & Muthen; 2004. Mplus. The comprehensive modeling program for applied researchers.
- [Background] Jöreskog KG, Sörbom D. LISREL 8.71 for Windows [computer program]. Lincolnwood, IL; Scientific Software International, Inc.; 2004.
- [Background] Karlson CW, Hamilton NA, Rapoff MA. Massage on experimental pain in healthy females: a randomized controlled trial. J Health Psychol. 2014 Mar;19(3):427-40. doi: 10.1177/1359105312471572. Epub 2013 Jan 29. PMID 23362336
- [Background] Maakaron, JE., Taher, AT. (2022). Sickle Cell Disease. Medscape. https://emedicine.medscape.com/article/205926-overview#showall
- [Background] U.S. Anti-Doping Agency. Nutrition Guide (2023). https://www.usada.org/athletes/substances/nutrition/fluids-and-hydration/
- [Background] Pinto DMR, do Sacramento MS, Santos PHS, Silva WS, de Oliveira EC, Gardenghi G, Ladeia AMT, Petto J. Physical exercise in sickle cell anemia: a systematic review. Hematol Transfus Cell Ther. 2021 Jul-Sep;43(3):324-331. doi: 10.1016/j.htct.2020.06.018. Epub 2020 Sep 15. PMID 33032952
- [Background] Scherr J, Wolfarth B, Christle JW, Pressler A, Wagenpfeil S, Halle M. Associations between Borg's rating of perceived exertion and physiological measures of exercise intensity. Eur J Appl Physiol. 2013 Jan;113(1):147-55. doi: 10.1007/s00421-012-2421-x. Epub 2012 May 22. PMID 22615009
- [Background] MacIntosh BR, Murias JM, Keir DA, Weir JM. What Is Moderate to Vigorous Exercise Intensity? Front Physiol. 2021 Sep 22;12:682233. doi: 10.3389/fphys.2021.682233. eCollection 2021. PMID 34630133
- [Background] Karlson CW, Barajas KG, Seals SR, Britt AB, Schlenz AM, Jackson EA, Davis DB, Morris MC, Valrie CR. Longitudinal Predictors of Pain in Pediatric Sickle Cell Disease. J Pediatr Psychol. 2023 Jul 5;48(6):553-561. doi: 10.1093/jpepsy/jsad017. PMID 37043758
- [Background] Marbrey, C., Davis, J., Morris, M., Jackson, E., & Karlson, C. Predictors of emergency department utilization and hospitalization for vaso-occlusive pain crises in pediatric patients with sickle cell disease. Pediatr Emerg Care Med Open Access. 2021 Jan:6(5):1-4